CLINICAL TRIAL: NCT07303062
Title: Evaluating the Impact of Adolescent Mental Health Parenting Program for Child-Adult Relationship Enhancement (AMP-CARE)
Brief Title: Adolescent Mental Health Parenting Program for Child-Adult Relationship Enhancement
Acronym: AMP-CARE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20-3652
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Adolescent Behavior
Keywords: teen parenting program; teen mental health; mental health stigma; positive parenting; parenting self-efficacy
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either intervention (AMP-CARE) or waitlist control
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AMP-CARE (Experimental): Parents will attend the 6 virtual sessions with a group of about 5-10 parents and 2 facilitators. The AMP-CARE group sessions are held for about 90 minutes once per week. Sessions include didactics, role playing, vignettes, and weekly home practice to build positive parenting techniques.
  Interventions: Behavioral: Adolescent Mental Health Parenting Program for Child-Adult Relationship Enhancement (AMP-CARE)
- Waitlist Control (No Intervention): Parents in the control group will be offered the intervention after completing the second study questionnaire.

INTERVENTIONS:
Behavioral: Adolescent Mental Health Parenting Program for Child-Adult Relationship Enhancement (AMP-CARE) — The goals of AMP-CARE are to teach parents how to form a positive relationship with their teen and to teach about typical adolescent development and mental health. Each AMP-CARE session will be led by 1 or 2 trainers. About 4 to 13 parents will attend each virtual session lasting approximately 1.5 hours. Sessions will be weekly for 6 weeks. Participants are encouraged to practice the skills learned at AMP-CARE between the sessions.
  Arms: AMP-CARE

SUMMARY:
The purpose of this research study is to learn if a parenting program called Adolescent Mental Health Parenting Program for Child Adult Relationship Enhancement (AMP-CARE) can help parents have more confidence in parenting their teen and improve their knowledge about normal teen development and teen mental health. The main questions it aims to answer are:

* Does the AMP-CARE parenting program improve confidence in teen parenting and positive parenting?
* Does the AMP-CARE parenting program improve parent knowledge about mental health?

Researchers will compare participants who complete the parenting program to those who do not.

Participants will:

* Complete 2 surveys, one at the start of the study and one 6 -12 weeks later
* Half of the participants will be randomly picked to attend the 6 virtual AMP-CARE sessions right away.
* The other half will have the opportunity to attend AMP-CARE after they complete the second survey.

DETAILED DESCRIPTION:
In this randomized controlled trial, 60 parents of teens, ages 11-14 years, will be randomized to either AMP-CARE or wait-list control to achieve the following aims:

AIM 1. To measure the impact of AMP-CARE on parent mental health literacy as measured by the Parental Child Mental Health Literacy Questionnaire (PCMHLQ).

AIM 2: To measure the impact of AMP-CARE on parenting self-efficacy as measured by the Parenting Self Efficacy Scale.

AIM 3: To measure the impact of AMP-CARE on promotive parenting practices assessed by the Positive Parenting and Parental Involvement subscales of the Alabama Parenting Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Parent or guardian of teen age 11-14 years
* Receiving primary care at selected study sites
* English speaking

Exclusion Criteria:

* Parents of children with severe mental illness (indicated by psychiatric hospitalization in the last 12 months or previous diagnosis of psychosis)
* Parents of children with severe developmental delay (indicated by prior diagnosis of severe neurodevelopmental impairment, global developmental delay, severe expressive language delay)
* Not available at time group is scheduled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Parent Mental Health Literacy | From enrollment to completion of AMP-CARE program or 6-12 weeks after enrollment.
  Parent Mental Health Literacy was assessed with 23-item self-report measure, the Parental Child Mental Health Literacy Questionnaire. Using a 5-pt scale with endpoints of "0=strongly disagree" and "4=strongly agree," parents were asked to indicate their level of agreement with statements related to 5 constructs: mental health recognition, beliefs, knowledge, help-seeking confidence, and fear of stigma. Scores ranged from 0 to 4. Higher scores indicate greater literacy.

SECONDARY OUTCOMES:
Parent Self Efficacy | From enrollment to completion of AMP-CARE program or 6-12 weeks after enrollment.
  Parenting self-efficacy was assessed with the 19-item self-report measure Parenting Self Efficacy Scale. Using a 5-point scale, parents indicated how frequently states related to their efficacy to develop positive teenager behavior, their efficacy to respond competently to negative teenager behavior, and their monitoring efficacy were true from "1=never" to 5 "always." Total scores ranged from 1 to 5 with higher scores indicating greater self-efficacy.
Promotive Parenting Practices | From enrollment to completion of AMP-CARE program or 6-12 weeks after enrollment.
  Promotive parenting practices were assessed with 16 self-report items from two subscales of Alabama Parenting Questionnaire. The positive involvement subscale includes 10 items, with a range of possible scores from 10 to 50. The positive parenting subscale includes 6 items, with a range of possible scores from 6 to 30. Parents rate the frequency with which each parenting practice occurs in their home from "1=never" to "5=always." Higher scores indicate more positive parenting.

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Schilling, MD MSHP, Study Director — University of North Carolina, Chapel Hill; Yasamin Sanii, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - UNC Pediatrics at Panther Creek, Cary, North Carolina
  - UNC Children's Primary and Specialty Care at Carolina Pointe II, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No